CLINICAL TRIAL: NCT00999388
Title: Shanghai Parkinson's Study
Status: Completed | Type: Observational
Sponsor: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999910001; 10-E-N001
Record Dates: First submitted 2009-10-20; First posted 2009-10-21 (Estimated); Last update posted 2018-04-05 (Actual); Status verified 2018-01-25

CONDITIONS: Parkinson's Disease
Keywords: Lifestyle; Environment; Neurodegenerative Diseases; Elderly; Public Health; PD; Parkinson Disease
MeSH Terms: conditions — Parkinson Disease; Neurodegenerative Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
Background:

* Parkinson disease (PD) is the second most prevalent neurodegenerative disease, affecting more than 1 percent of the elderly population in the United States and other Western countries. Although effective treatments can alleviate symptoms in early PD, no cure or treatment slowing disease progression has been identified, and patients will eventually develop severe physical and mental disabilities and often die of complications. More research is needed on the causes of and appropriate preventive strategies for PD.
* The Shanghai Women s Health Study (SWHS) was established 10 years ago by investigators from the Vanderbilt University, the Shanghai Cancer Institute (SCI) and the National Cancer Institute (NCI) of the US. Their primary aim was to examine several unique dietary hypotheses on cancer among Chinese women. Researchers from the National Institute of Environmental Health Sciences and SWHS investigators are now interested in studying PD patients from SWHS to evaluate biological and environmental factors that may have put them at risk for PD.

Objectives:

* To initiate a long-term prospective study on PD in Chinese women from the Shanghai Women s Health Study.
* To examine a set of biological and environmental factors that may raise or lower risk of developing PD.

Eligibility:

- All participants of the SWHS cohort are eligible.

Design:

* Researchers will contact self-reported PD cases from the SWHS, confirm (or reject) the self-report, and invite them to a clinical examination at a coordinating hospital in Shanghai.
* Cases that confirm the self-report will be invited to visit the coordinating hospital for clinical examinations, including a PD clinical workup, blood and urine collections, a cognitive assessment and relevant neuropsychological testing, and an interview on additional risk factor exposures that are not available from baseline surveys.
* For those who could not participate in the clinical examination, researchers will ask for a few details about the diagnosis and treatment history and ask for permission to obtain medical records relevant to PD diagnosis from government or hospital agencies.
* For self-reported PD cases who are now deceased, researchers will follow a similar procedure by asking for consent and help from the next-of-kin.

DETAILED DESCRIPTION:
We propose to clinically examine self-reported Parkinson s disease (PD) patients from the well established Shanghai Women s Health Study (SWHS) and thus initiate a long-term PD research in this unique Chinese women cohort. The SWHS cohort was established in late 1990s by Dr. Wei Zheng from Vanderbilt University in collaboration with investigators from the Shanghai Cancer Institute (SCI) and the National Cancer Institute (NCI) of the US. Their primary aim was to examine several unique dietary hypotheses on cancer among Chinese women. From 1996 to 2000, the SWHS successfully recruited 74,942 Chinese women, aged 40 to 70, from selected communities in a single district in Shanghai with an overall consent rate of 92%. All participants completed a comprehensive baseline survey, 88% donated urine, 76% donated blood, and an additional 12% donated buccal cells.1 Follow-up surveys have since been conducted biennially with consistent participation rates of 95% or higher. Through the 3rd follow-up, the cohort has documented 220 self-reported PD cases and we expect to identify another 80 self-reports during the ongoing 4th follow-up survey (2007-2010). We hereby propose to clinically examine self-reported PD patients to achieve the following two major aims.

Aim #1: To initiate a long-term prospective study on PD in this unique Chinese women cohort

Aim #2: To examine the following specific hypotheses among women

1. <TAB>Higher plasma levels of pro-inflammatory biomarkers predict higher PD risk.
2. <TAB>Higher plasma uric acid is associated with a lower PD risk
3. <TAB>Environmental tobacco smoke (ETS) is associated with lower PD risk

   1. Self-reported ETS exposure is associated with a lower PD risk
   2. Higher urine level of cotinine is associated with a lower PD risk

We hereby propose a prospective study on PD in a unique women-only cohort. The infrastructure and the many desirable characteristics of this cohort offer us a rare opportunity for PD research in women, particularly on biomarkers. We expect to establish it as a long-term and excellent resource for PD research in women in the future. In the short term, we plan to examine several promising PD hypotheses that have not been adequately evaluated among women. These findings will apply directly to Chinese women and may also have implications for women in the West. PD etiological research is under-represented in women. Therefore, research in the SPS may not only corroborate findings on women in the west, but also lead to the identification of novel risk factors that could be generalizable to Western women.

ELIGIBILITY:
* Inclusion and exclusion criteria:

This study will be conducted within the infrastructure of the Shanghai Women s Health Study. At this stage, all self-reported PD cases through the 4th follow-up will be invited. As the 4th follow-up is ongoing, we will start with cases identified from the first three follow-ups and add new cases as they are identified. Through the 3rd follow-up, a total of 220 PD patients have self-identified and 141 are incident. Assuming 200 cases are still alive at the time of the proposed study and another 80 are self-identified during the 4th follow-up, we will have approximately 280 self-reported PD patients that are eligible for the clinical confirmation at current stage. Cases identified from future SWHS follow-ups will be eligible for future SPS work.

Analyses on biomarkers and genes will be conducted in a case-control manner. Overall, two controls will be selected for each case, individually matched on year of birth (+/-1), and maybe some other factors such as survival status, baseline menopausal status, fasting status, season of specimen collection, and time of the day of specimen collection. These controls have provided exposure data and/or biospecimen at baseline. Therefore at current stage no active field data collection will be carried out for controls.

As at the current stage, the expected number of Parkinson cases is small, therefore we do not plan to pre-exclude any participants from this study.

Ages: 40 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 149 (Actual)
Dates: Start 2009-10-14; Study Completion 2018-01-25

PRIMARY OUTCOMES:
A long-term prospective study of PD in this cohort | Ongoing

CONTACTS AND LOCATIONS:
Overall Officials: Gitanjali Taneja, Ph.D., Principal Investigator — National Institute of Environmental Health Sciences (NIEHS)
Locations (2):
- China (2):
  - Fudan University Huashan Hospital Shanghai, Shanghai
  - Shanghai Cancer Institute, Shanghai

REFERENCES:
- [Background] Gasser T. Genetics of Parkinson's disease. Curr Opin Neurol. 2005 Aug;18(4):363-9. doi: 10.1097/01.wco.0000170951.08924.3d. PMID 16003110
- [Background] Tanner CM, Ottman R, Goldman SM, Ellenberg J, Chan P, Mayeux R, Langston JW. Parkinson disease in twins: an etiologic study. JAMA. 1999 Jan 27;281(4):341-6. doi: 10.1001/jama.281.4.341. PMID 9929087
- [Background] Hernan MA, Takkouche B, Caamano-Isorna F, Gestal-Otero JJ. A meta-analysis of coffee drinking, cigarette smoking, and the risk of Parkinson's disease. Ann Neurol. 2002 Sep;52(3):276-84. doi: 10.1002/ana.10277. PMID 12205639